CLINICAL TRIAL: NCT05561738
Title: Nicotinamide Riboside in Ulcerative Colitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Crohn's and Colitis Foundation (Other)
Responsible Party: Principal Investigator, Kevin Mollen, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: STUDY22060104
Record Dates: First submitted 2022-09-13; First posted 2022-09-30 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis
Keywords: NAD
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Daily oral therapy with Nicotinamide Riboside Chloride (Niagen) + Standard Therapy (Experimental): Nicotinamide Riboside Chloride (Niagen) 75mg or 250mg capsules provided by ChromaDex, Inc. Dosing is recommended at 12.5mg/kg/day.
  The dosing plan is as follows (in mg po qD):
  20-25 kg 250mg; 25-30 kg 325mg; 30-35 kg 400mg; 35-40 kg 475mg; 40-45 kg 500mg; 45-50 kg 575mg; 50-55 kg 650mg; 55-60 kg 725mg; 60-65 kg 750mg; 65-70 kg 825mg; >70 kg 900mg (max dosing).
  Interventions: Dietary Supplement: Nicotinamide Riboside Chloride; Other: Standard of Care
- Daily oral therapy with placebo + Standard Therapy (Experimental): Placebo 75mg or 250mg capsules provided by ChromaDex, Inc. Dosing is recommended at 12.5mg/kg/day.
  The dosing plan is as follows (in mg po qD):
  20-25 kg 250mg; 25-30 kg 325mg; 30-35 kg 400mg; 35-40 kg 475mg; 40-45 kg 500mg; 45-50 kg 575mg; 50-55 kg 650mg; 55-60 kg 725mg; 60-65 kg 750mg; 65-70 kg 825mg; >70 kg 900mg (max dosing).
  Interventions: Dietary Supplement: Placebo; Other: Standard of Care

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside Chloride — The intervention consists of 6 months to 1 year of daily oral therapy with Nicotinamide Riboside Chloride (Niagen) in addition to standard therapy.
  Arms: Daily oral therapy with Nicotinamide Riboside Chloride (Niagen) + Standard Therapy
Dietary Supplement: Placebo — The intervention consists of 6 months to 1 year of daily oral therapy with placebo (Maltodextran capsules of similar size, shape and color as Niagen) in addition to standard therapy.
  Arms: Daily oral therapy with placebo + Standard Therapy
Other: Standard of Care — Standard of Care

SUMMARY:
This is a randomized, double-blind pilot study of Nicotinamide Riboside (NR) in Pediatric-onset Ulcerative Colitis (UC).

DETAILED DESCRIPTION:
The investigators hypothesize that NR will alleviate mitochondrial dysfunction and restore metabolic homeostasis in the intestinal epithelium in pediatric patients with UC.

The purpose of the study are:

1. To establish the feasibility of an Randomized Clinical Trial (RCT) investigating the effects of NR in pediatric patients with UC.
2. To evaluate the effects of Nicotinamide adenine dinucleotide (NAD)+ repletion on intestinal epithelial mitochondrial structure and function in human UC patients. The investigators hypothesize that daily NR supplementation will restore NAD+ levels, enhancing Peroxisome proliferator-activated receptor gamma coactivator 1-alpha (PGC1α) activity and mitochondrial structure/function.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (≤18yo);
* Diagnosis of mild to moderate ulcerative colitis as determined by Pediatric Ulcerative Colitis Activity Index (PUCAI) and endoscopic scoring (Mayo) at the time of colonoscopy;
* Although the investigators will target newly diagnosed patients (therefore, treatment naïve), patients with established disease will also be enrolled.

Exclusion Criteria:

* Patients with acute severe ulcerative colitis;
* Concurrent gastrointestinal infection (ie. Clostridium difficile, Cytomegalovirus, etc.);
* A diagnosis of Crohn's disease;
* Indeterminate colitis/IBD-U;
* In general, patients that have been treated with steroids or antibiotics in the past three months. Patients on Biologic medications may be enrolled if their dose has been stable for at least three months. Final determination of eligibility will be at the discretion of the treating investigator. After the initiation of the study, subjects may receive any medication to treat their disease as dictated by their care providers;
* Patients who have other chronic inflammatory/autoimmune disorders or prior malignancy;
* Pregnant women (All women of childbearing age will be required to use contraception at the time of inclusion).
* Patients with existing renal or hepatic dysfunction;
* Per standard of care guidance, subjects with platelets <50,000 do not undergo endoscopy and, therefore, are not eligible.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients screened | 2 years
  The investigators will report the number of overall patients screened for enrollment.
Proportion of patients screened who meet inclusion/exclusion criteria | 2 years
  The investigators will report the number of patients screened who meet inclusion/exclusion criteria.
Enrollment percentage | 2 years
  The investigators will report the proportion of eligible patients who enroll in the study per month.
Completion percentage | 2 years
  The investigators will report the proportion of enrolled subjects who complete the study.
Reasons for exclusion | 2 years
  The investigators will report the reasons that patients are excluded from the study.
Dropout rate | 2 years
  The investigators will report the percentage of subjects who drop out per month.
Reasons for dropout | 2 years
  The investigators will log reasons for dropout.

SECONDARY OUTCOMES:
Changes in mitochondrial structure from baseline to 6-12 months | Baseline 6-12 months
  Subjects will undergo colonoscopic evaluation at enrollment and after 6-12 months of treatment (per standard treatment protocols). Investigators will perform a qualitative analysis of mitochondrial structure using scanning electron microscopy and/or immunofluorescence at both timepoints.
Changes in mitochondrial function from baseline to 6-12 months | Baseline 6-12 months
  Subjects will undergo colonoscopic evaluation at enrollment and after 6-12 months of treatment (per standard treatment protocols). Investigators will evaluate mitochondrial function (Complex 1 and 2) via the Oroboros 2K Analyzer [oxygen consumption [(pmol/(s × mL)/μg protein] at both timepoints.
Changes in the PGC1α-Sirt1 axis from baseline to 6-12 months | Baseline 6-12 months
  Subjects will undergo colonoscopic evaluation at enrollment and after 6-12 months of treatment (per standard treatment protocols). PGC1α and Sirt1 levels will be evaluated in tissue biopsies using western blot (qualitative analysis of protein levels) and qRT-PCR analysis (quantitative gene expression in fold change) at both timepoints.
Changes in cellular metabolism from baseline to 6-12 months | Baseline 6-12 months
  Subjects will undergo colonoscopic evaluation at enrollment and after 6-12 months of treatment (per standard treatment protocols). An untargeted metabolomic analysis of the intestinal epithelium will be performed at these time points (fold change) at both timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Mollen, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data and samples may be shared with the funding agent, other researchers or federal repositories in the future under and approved agreement.
Supporting Information: Study Protocol, CSR
Time Frame: 6 months after publication of the results of the study. Date will be available for 1 year.
Access Criteria: Prior to any sharing of any data, the research data/documents will be coded and all subject identifiers will be completely removed. Only the PI and co-investigators will have access to the coding. All others will have access to the completely deidentified data only.
  A data use agreement will be obtained and finalized prior to any of the data leaving the institution, and prior to any access by outside entities.

REFERENCES:
- [Background] Novak EA, Mollen KP. Mitochondrial dysfunction in inflammatory bowel disease. Front Cell Dev Biol. 2015 Oct 1;3:62. doi: 10.3389/fcell.2015.00062. eCollection 2015. PMID 26484345
- [Background] Cunningham KE, Vincent G, Sodhi CP, Novak EA, Ranganathan S, Egan CE, Stolz DB, Rogers MB, Firek B, Morowitz MJ, Gittes GK, Zuckerbraun BS, Hackam DJ, Mollen KP. Peroxisome Proliferator-activated Receptor-gamma Coactivator 1-alpha (PGC1alpha) Protects against Experimental Murine Colitis. J Biol Chem. 2016 May 6;291(19):10184-200. doi: 10.1074/jbc.M115.688812. Epub 2016 Mar 11. PMID 26969166
- [Background] Haberman Y, Karns R, Dexheimer PJ, Schirmer M, Somekh J, Jurickova I, Braun T, Novak E, Bauman L, Collins MH, Mo A, Rosen MJ, Bonkowski E, Gotman N, Marquis A, Nistel M, Rufo PA, Baker SS, Sauer CG, Markowitz J, Pfefferkorn MD, Rosh JR, Boyle BM, Mack DR, Baldassano RN, Shah S, Leleiko NS, Heyman MB, Grifiths AM, Patel AS, Noe JD, Aronow BJ, Kugathasan S, Walters TD, Gibson G, Thomas SD, Mollen K, Shen-Orr S, Huttenhower C, Xavier RJ, Hyams JS, Denson LA. Ulcerative colitis mucosal transcriptomes reveal mitochondriopathy and personalized mechanisms underlying disease severity and treatment response. Nat Commun. 2019 Jan 3;10(1):38. doi: 10.1038/s41467-018-07841-3. PMID 30604764
- [Background] Larmonier CB, Shehab KW, Laubitz D, Jamwal DR, Ghishan FK, Kiela PR. Transcriptional Reprogramming and Resistance to Colonic Mucosal Injury in Poly(ADP-ribose) Polymerase 1 (PARP1)-deficient Mice. J Biol Chem. 2016 Apr 22;291(17):8918-30. doi: 10.1074/jbc.M116.714386. Epub 2016 Feb 24. PMID 26912654
- [Background] Santos L, Escande C, Denicola A. Potential Modulation of Sirtuins by Oxidative Stress. Oxid Med Cell Longev. 2016;2016:9831825. doi: 10.1155/2016/9831825. Epub 2015 Dec 14. PMID 26788256
- [Background] Gerner RR, Klepsch V, Macheiner S, Arnhard K, Adolph TE, Grander C, Wieser V, Pfister A, Moser P, Hermann-Kleiter N, Baier G, Oberacher H, Tilg H, Moschen AR. NAD metabolism fuels human and mouse intestinal inflammation. Gut. 2018 Oct;67(10):1813-1823. doi: 10.1136/gutjnl-2017-314241. Epub 2017 Sep 6. PMID 28877980
- [Background] Mehmel M, Jovanovic N, Spitz U. Nicotinamide Riboside-The Current State of Research and Therapeutic Uses. Nutrients. 2020 May 31;12(6):1616. doi: 10.3390/nu12061616. PMID 32486488
- [Background] Trammell SA, Schmidt MS, Weidemann BJ, Redpath P, Jaksch F, Dellinger RW, Li Z, Abel ED, Migaud ME, Brenner C. Nicotinamide riboside is uniquely and orally bioavailable in mice and humans. Nat Commun. 2016 Oct 10;7:12948. doi: 10.1038/ncomms12948. PMID 27721479
- [Background] Jiang Y , Liu Y , Gao M , Xue M , Wang Z , Liang H . Nicotinamide riboside alleviates alcohol-induced depression-like behaviours in C57BL/6J mice by altering the intestinal microbiota associated with microglial activation and BDNF expression. Food Funct. 2020 Jan 29;11(1):378-391. doi: 10.1039/c9fo01780a. PMID 31820774